CLINICAL TRIAL: NCT07204119
Title: Official Title: Comparison of Graston Technique With Tissue Flossing Technique in Patient With Post-Operative Knee Stiffness
Brief Title: Comparison of GT With TF Technique in Patient With Post-Operative Knee Stiffness
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Riphah/RCRS/REC/02181
Record Dates: First submitted 2025-09-25; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Post-operative Knee Stiffness
Keywords: Post-operative knee stiffness; Graston Technique; Range of Motion; Tissue Flossing
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tissue Flossing Technique (Experimental): Hot pack: 10 minutes, PNF (hold-relax with agonist contraction), CPM: 10 minutes, Self-stretching: End range position for 30 seconds, repeat twice.
  1 to 2 minutes for Tissue Flossing Technique Description: Active and passive movement with knee wrapped in a high-quality floss band (208×5×0.15 cm), Wrapped from upper gastrocnemius to lower quadriceps and hamstring muscles using a 50% overlapping pattern with a 25% elongation stretch, Series of active and passive exercises (knee flexion and extension) with 3 repetitions.
  Interventions: Other: Tissue Flossing Technique
- Graston Technique (Experimental): Hot pack: 10 minutes, PNF (hold-relax with agonist contraction), CPM: 10 minutes, Self-stretching: End range position for 30 seconds, repeat twice.
  2 minutes for Graston Technique Technique Description: Participant lies supine with hip and knee straight, Water-based gel used to reduce friction.
  Superior and inferior longitudinal strokes delivered with GT-4 instrument at a 45° angle to soft tissues Sequence includes strokes from above patella to anterior inferior iliac spine (AIIS) and back, maintaining a 2-second cadence
  Interventions: Other: Graston Technique
- Control group (Active Comparator): Hot pack: 10 minutes
  * PNF (hold-relax with agonist contraction): Gentle stretch of knee muscle for 10 seconds Isometric contraction for 6 seconds. Flex knee with therapist assistance. Hold position for 10 seconds, repeat 3 times
  * CPM: 10 minutes
  * Self-stretching: End range position for 30 seconds, repeat twice
  Interventions: Other: Control group

INTERVENTIONS:
Other: Tissue Flossing Technique — Hot pack: 10 minutes, PNF (hold-relax with agonist contraction), CPM: 10 minutes, Self-stretching: End range position for 30 seconds, repeat twice. 1 to 2 minutes for Tissue Flossing Technique Description: Active and passive movement with knee wrapped in a high-quality floss band (208×5×0.15 cm), Wrapped from upper gastrocnemius to lower quadriceps and hamstring muscles using a 50% overlapping pattern with a 25% elongation stretch, Series of active and passive exercises (knee flexion and extension) with 3 repetitions.
  Arms: Tissue Flossing Technique
Other: Graston Technique — Hot pack: 10 minutes, PNF (hold-relax with agonist contraction), CPM: 10 minutes, Self-stretching: End range position for 30 seconds, repeat twice.
  2 minutes for Graston Technique Technique Description: Participant lies supine with hip and knee straight, Water-based gel used to reduce friction.
  Superior and inferior longitudinal strokes delivered with GT-4 instrument at a 45° angle to soft tissues Sequence includes strokes from above patella to anterior inferior iliac spine (AIIS) and back, maintaining a 2-second cadence
  Arms: Graston Technique
Other: Control group — Hot pack: 10 minutes, PNF (hold-relax with agonist contraction): Gentle stretch of knee muscle for 10 seconds Isometric contraction for 6 seconds. Flex knee with therapist assistance. Hold position for 10 seconds, repeat 3 times, CPM: 10 minutes, Self-stretching: End range position for 30 seconds, repeat twice
  Arms: Control group

SUMMARY:
The purpose of this study was to compare the effects of Graston Technique and Tissue Flossing Technique in patients with post-operative knee stiffness on pain, range of motion, and functional outcomes. A randomized controlled trial was conducted at Benazir Bhutto Hospital, Rawalpindi. The total sample size was 48, divided into three groups. The study duration was six months. Purposive sampling was applied for recruitment, and group randomization was performed by lottery method. Only patients with post-operative knee stiffness meeting the inclusion criteria were enrolled. Outcome measures included goniometer, Functional Independence Measure (FIM), and Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) questionnaires. Data was collected at baseline and after interventions, and analysis was performed using SPSS version 23.

DETAILED DESCRIPTION:
Stiffness has been defined as a decrease in postoperative range of motion (ROM), including flexion contracture, accompanied by persistent pain and/or functional compromise (1). Post-traumatic stiffness may result from dense intra-articular adhesions and fibrotic transformation of periarticular structures (2). The knee joint, crucial for lower-limb biomechanics, is the most frequently injured joint in the lower extremities (3). Post-traumatic knee stiffness and loss of ROM are common complications following knee injuries. The normal ROM of the knee joint is generally accepted to be 0° (full extension) to 135° (full flexion). A stiff knee is defined as one with a total ROM of less than 50°, while an ankylosed knee is characterized by a ROM of less than 30° (4). Knee joint stiffness may result from several factors, including periarticular surgeries, traumatic injuries, inflammatory or infectious joint diseases, fractures, prolonged immobilization, and scar formation due to burns or trauma. Post-surgical procedures such as open reduction and internal fixation (ORIF) may also contribute to stiffness through scar tissue formation and reduced joint mobility (5). The choice of fixation method for femoral or tibial fractures depends on the fracture type and anatomical location. For femoral shaft fractures, intramedullary (IM) nailing is considered the gold standard. Stabilization of femoral or tibial fractures can also be achieved through ORIF using screws, plates, or rods. In cases with compromised skin integrity at the fracture site, external fixation provides a temporary solution, using external frames to align the bones (6) Diagnosis of post-operative knee stiffness is based on reduced knee flexion and extension after surgery, commonly following ORIF of femur, tibia, or fibula fractures. Literature defines stiffness as total knee ROM <50° and ankylosis when <30°. Clinical judgment with goniometric assessment and functional evaluation using WOMAC and FIM questionnaires provides valid measures. Previous studies suggest intra-articular adhesions, fibrotic changes, and prolonged immobilization as primary contributors to post-operative knee stiffness.

Various therapeutic interventions have been developed to address this issue, myofascial compression technique, i.e., Graston Technique and tissue flossing emerging as promising approaches. The Graston Technique (GT) is a therapeutic approach known as instrument-assisted soft tissue mobilization (IASTM). GT uses specialized tools to massage and scrape the skin, reducing pain and targeting tissue restrictions that cause dysfunction. The Graston Technique supports soft tissue healing by enhancing blood flow (vasodilation) to the affected area, which can accelerate recovery and reduce stiffness (7).

The Graston Technique, instrument-assisted soft tissue mobilization (IASTM), has shown efficacy in improving range of motion and reducing pain in various musculoskeletal conditions. Studies have demonstrated its effectiveness in treating chronic low back pain, with significant improvements in pain reduction and increased range of motion compared to general exercise alone (8).

The technique has also been found to be beneficial in addressing postoperative elbow stiffness, showing greater improvements in pain reduction and patient-specific function compared to other soft tissue mobilization techniques (9)

. For instance, a study on patients with anterior knee pain found that IASTM techniques, including the Graston Technique, were as effective as stretching exercises in reducing pain, improving flexibility, and enhancing lower extremity function in patients with iliotibial band tightness (10).

Similarly, compressive myofascial release techniques have demonstrated effectiveness in increasing ankle dorsiflexion range of motion (11).

Tissue flossing, on the other hand, utilizes a floss band that is elastic rubber band designed to wrap around joints or muscle groups before or during exercise or stretching. The primary mechanism involves blood flow restriction (BFR), creating temporary tissue ischemia, followed by blood flow reperfusion upon removal, which can boost metabolic responses (3).

Tissue flossing is a novel technique gaining popularity in athletic training and rehabilitation for its potential effects on joint range of motion (ROM) and muscle function. Studies have shown that floss band application on limbs, soft tissues, or joints with approximately 50% tension wrapping pressure can have small to medium effects on ROM, muscle stiffness, and strength (12).

Research on the effects of tissue flossing on joint stiffness has produced mixed results. Some studies have reported positive outcomes, such as increased ankle ROM and improved jump and sprint performance in recreational athletes (13).

The Graston Technique and tissue flossing are two techniques that aim to improve soft tissue mobility and joint function through distinct mechanisms. The former employs specialized instruments for soft tissue mobilization, while the latter uses compression and subsequent modulation of blood flow.

The lack of direct comparisons between these techniques underscores the potential significance of study investigating their comparative efficacy in treating post-operative knee stiffness. Such research could substantially contribute to the existing body of knowledge regarding soft tissue mobilization techniques and their applications across various musculoskeletal conditions, thereby providing clinicians with valuable insights.

ELIGIBILITY:
Inclusion Criteria:

1. Age group between 20 to 40 years.
2. Both male and female.
3. Patients with 6 weeks post-operative following open reduction and internal fixation (ORIF) of femur, tibia, or fibula shaft fracture
4. Decreased in knee Flexion & Extension (A minimum of 20° or above).

Exclusion criteria:

1. Those patients who have allergies to latex
2. Malignant or metabolic cause of knee fracture
3. Venous Thrombotic disease/ Varicose veins.
4. Cardiopulmonary illness and hypertension.
5. Skin diseases/ metabolic disorders.
6. Patient with arthroplasty and arthroscopy.
7. Patellar fracture/ ACL/ PCL/ MCL/ LCL rupture/ injuries.
8. Any pathological condition having effects on knees.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-02-12 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-25 (Estimated)

PRIMARY OUTCOMES:
Range of Motion: | 2 weeks
  Range of motion (ROM) is the extent of movement possible at a joint or body part. It's the arc of motion a joint can travel, typically measured in degrees using a goniometer. Healthy ROM allows for comfortable movement, while limitations can lead to pain and reduced function.

SECONDARY OUTCOMES:
Numerated Pain Rating Scale: | 2 weeks
  The Numeric Rating Scale (NRS), also known as the Numeric Pain Rating Scale (NPRS), is a simple, validated tool used to measure pain intensity by having a person rate their pain on a scale, typically from 0 to 10, where 0 means no pain and 10 means the worst possible pain.
Western Ontario and McMaster Universities Osteoarthritis Index | 2 weeks
  WOMAC stands for the Western Ontario and McMaster Universities Osteoarthritis Index, a self-administered questionnaire used by health professionals to assess osteoarthritis (OA) of the hip and knee. It measures pain, stiffness, and physical function through 24 items across three subscales, with higher scores indicating increased difficulty.
Functional Independence Measure: | 2 weeks
  The Functional Independence Measure (FIM) is an assessment tool used in rehabilitation to evaluate a patient's ability to perform daily activities by measuring the degree of assistance required.

CONTACTS AND LOCATIONS:
Overall Officials: Lal Gul Khan, MS, Principal Investigator — Riphah International University
Locations (1):
- Banazir Bhutto Hospital,, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Manrique J, Gomez MM, Parvizi J. Stiffness after total knee arthroplasty. J Knee Surg. 2015 Apr;28(2):119-26. doi: 10.1055/s-0034-1396079. Epub 2014 Dec 16. PMID 25513992
- [Background] Galvez-Sirvent E, Ibarzabal-Gil A, Rodriguez-Merchan EC. Complications of the surgical treatment of fractures of the tibial plateau: prevalence, causes, and management. EFORT Open Rev. 2022 Aug 4;7(8):554-568. doi: 10.1530/EOR-22-0004. PMID 35924649
- [Background] Wu SY, Tsai YH, Wang YT, Chang WD, Lee CL, Kuo CA, Chang NJ. Acute Effects of Tissue Flossing Coupled with Functional Movements on Knee Range of Motion, Static Balance, in Single-Leg Hop Distance, and Landing Stabilization Performance in Female College Students. Int J Environ Res Public Health. 2022 Jan 27;19(3):1427. doi: 10.3390/ijerph19031427. PMID 35162447
- [Background] Pirato F, Rosso F, Dettoni F, Bonasia DE, Bruzzone M, Rossi R. How to manage a native stiff knee. EFORT Open Rev. 2024 May 10;9(5):363-374. doi: 10.1530/EOR-24-0034. PMID 38726987
- [Background] Phruetthiphat OA, Zampogna B, Vasta S, Tassanawipas B, Gao Y, Callaghan JJ. TKR after posttraumatic and primary knee osteoarthritis: a comparative study. J Orthop Surg Res. 2021 Mar 4;16(1):173. doi: 10.1186/s13018-021-02322-8. PMID 33663576
- [Background] Mckivigan JM, Tulimero G. An Analysis Of Graston Technique® For Soft-Tissue Therapy. Rehabilitation Science. 2020;5(4):31. 2020.
- [Background] 26, Kangra Rm. Effectiveness Of Instrument Assisted Soft Tissue Mobilization (Iastm) On Post-Operative Knee Stiffness: A Case Study. International Journal Of Scientific Research. 2024 Jun; 13(5).
- [Background] Lee JH, Lee DK, Oh JS. The effect of Graston technique on the pain and range of motion in patients with chronic low back pain. J Phys Ther Sci. 2016 Jun;28(6):1852-5. doi: 10.1589/jpts.28.1852. Epub 2016 Jun 28. PMID 27390432
- [Background] Bhosale P, Kolke Pt S. Effectiveness of instrument assisted soft tissue mobilization (IASTM) and muscle energy technique (MET) on post-operative elbow stiffness: a randomized clinical trial. J Man Manip Ther. 2023 Oct;31(5):340-348. doi: 10.1080/10669817.2022.2122372. Epub 2022 Sep 28. PMID 36171728
- [Background] Lim, J.-Y., Nam, S.-H., & Kim, K.-D. (2022). Effect of Active Stretching and Instrument-Assisted Soft Tissue Mobilization on the Hip Joint Range of Motion and Stiffness of the Tensor Fascia Lata in Subjects with Shortened Tensor Fascia Lata. Journal of Musculoskeletal Science and Technology, 6(2), 43-50.
- [Background] Stanek J, Sullivan T, Davis S. Comparison of Compressive Myofascial Release and the Graston Technique for Improving Ankle-Dorsiflexion Range of Motion. J Athl Train. 2018 Feb;53(2):160-167. doi: 10.4085/1062-6050-386-16. Epub 2018 Jan 26. PMID 29373060
- [Background] Jianhong, G., Seng, T. J., Samsudin, S., Soon, C. C., & Zaremohzzabieh, Z. (2021). The Effect of Tissue Flossing Technique on Sports and Injury Prevention and Rehabilitation: A Systematic Review of Recent Research. International Journal of Human Movement and Sports Sciences, 9(6), 1157-1173.
- [Background] Mills B, Mayo B, Tavares F, Driller M. The Effect of Tissue Flossing on Ankle Range of Motion, Jump, and Sprint Performance in Elite Rugby Union Athletes. J Sport Rehabil. 2020 Mar 1;29(3):282-286. doi: 10.1123/jsr.2018-0302. PMID 30676229
- [Background] Cheatham SW, Kolber MJ, Mokha M, Hanney WJ. Concurrent validity of pain scales in individuals with myofascial pain and fibromyalgia. J Bodyw Mov Ther. 2018 Apr;22(2):355-360. doi: 10.1016/j.jbmt.2017.04.009. Epub 2017 Apr 27. PMID 29861234
- [Background] Hancock GE, Hepworth T, Wembridge K. Accuracy and reliability of knee goniometry methods. J Exp Orthop. 2018 Oct 19;5(1):46. doi: 10.1186/s40634-018-0161-5. PMID 30341552
- [Background] Danish M, Thakare AE, Salkar PS, Wakode SL. Clinical Utility of Blood Pressure Measurement Using the Newer Palpatory Method for Both Systolic and Diastolic Blood Pressure. Adv Biomed Res. 2020 Sep 30;9:51. doi: 10.4103/abr.abr_254_19. eCollection 2020. PMID 33457334
- [Background] Impellizzeri FM, Mannion AF, Leunig M, Bizzini M, Naal FD. Comparison of the reliability, responsiveness, and construct validity of 4 different questionnaires for evaluating outcomes after total knee arthroplasty. J Arthroplasty. 2011 Sep;26(6):861-9. doi: 10.1016/j.arth.2010.07.027. Epub 2010 Nov 12. PMID 21074964
- [Background] Gkouma A, Theotokatos G, Geladas N. Validity and Reliability Evidence of the Functional Independence Measurement (FIM) for individuals with Neurological Disorders in Greece. J Med-Clin Res & Rev. 2022;6(5):1-1.